CLINICAL TRIAL: NCT04375852
Title: Tyrosine Hydroxylase Antibody Levels in Autoimmune Polyglandular Syndrome Type 1 Associated Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TEC 2020-001
Record Dates: First submitted 2020-04-26; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Autoimmune Polyglandular Syndrome Type I; Autoimmune Keratitis
Keywords: Tyrosine hydroxylase; Autoantibodies; Autoimmune Polyglandular Syndrome
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): consecutive cases diagnosed with APS-1associated keratitis
  Interventions: Diagnostic Test: Detection of autoantibodies

INTERVENTIONS:
Diagnostic Test: Detection of autoantibodies — Blood was obtained from each patient for testing the endocrine functions and determination of a panel of autoantibodies to the following: Side-chain cleavage enzyme (SSC), Aromatic L-amino acid decarboxylase (AADC), Tryptophan hydroxylase (TPH),Tyrosine hydroxylase ( TH), 17α-hydroxylase (17α-OH), Cytochrome P450 1A2 (CYP1A2), 21-hydroxylase (21-OH), Potassium channel regulatory protein (KCNRG), Tyrosine phosphatase-like protein IA-2 (IA-2), Glutamic acid decarboxylase 65 (GAD65), NACT Leucine-Rich-Repeat-Protein 5 (NALP5), and Interleukin (IL) 22.

SUMMARY:
Tyrosine hydroxylase autoantibodies impair sympathetic innervation leading to keratitis. In this study, the investigators have shown the significant association between severity of keratitis and presence of tyrosine hydroxylase autoantibodies.

DETAILED DESCRIPTION:
Sixteen consecutive cases diagnosed with APS-1associated keratitis were included in this study. Each patient underwent complete ophthalmologic examination. Blood was obtained from each patient for testing the endocrine functions and determination of a panel of autoantibodies to the following: Side-chain cleavage enzyme (SSC), Aromatic L-amino acid decarboxylase (AADC), Tryptophan hydroxylase (TPH),Tyrosine hydroxylase ( TH), 17 α-hydroxylase (17α-OH), Cytochrome P450 1A2 (CYP1A2), 21-hydroxylase (21-OH), Potassium channel regulatory protein (KCNRG), Tyrosine phosphatase-like protein IA-2 (IA-2), Glutamic acid decarboxylase 65 (GAD65), NACT Leucine-Rich-Repeat-Protein 5 (NALP5), and Interleukin (IL) 22.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients diagnosed with APS-1associated keratitis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

PRIMARY OUTCOMES:
To report the correlation between autoantibodies with the severity keratitis in patients Autoimmune polyglandular syndrome type 1 (APS-1). | 3 months
  Blood was obtained from each patient for determination of a panel of autoantibodies to the following: Side-chain cleavage enzyme (SSC), Aromatic L-amino acid decarboxylase (AADC), Tryptophan hydroxylase (TPH),Tyrosine hydroxylase ( TH), 17α-hydroxylase (17α-OH), Cytochrome P450 1A2 (CYP1A2), 21-hydroxylase (21-OH), Potassium channel regulatory protein (KCNRG), Tyrosine phosphatase-like protein IA-2 (IA-2), Glutamic acid decarboxylase 65 (GAD65), NACT Leucine-Rich-Repeat-Protein 5 (NALP5), and Interleukin (IL) 22.

IPD SHARING:
Plan to Share IPD: No